CLINICAL TRIAL: NCT06805760
Title: Ventilation Strategies Impact on Oxygenation and Postoperative Pulmonary Complications in Lung Surgery Patients: a Prospective, Randomized, Triple-Blind Trial
Brief Title: Ventilation Strategies Impact on Oxygenation and Postoperative Pulmonary Complications in Lung Surgery Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inner Mongolia Baogang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024-MER-313
Record Dates: First submitted 2025-01-20; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Lung Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- V-VCV Group (Experimental): The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW).The maximum tidal volume (Vt_max) and minimum tidal volume (Vt_min) were set at 10-20% of the basal tidal volume (Vt_base). Respiratory Rate 12. Inspiratory Flow Rate (IFR) 60L/min, Inspiratory to Expiratory Ratio (IER) 1:2, Positive End-Expiratory Pressure (PEEP) 5cm water column, and Inhaled Oxygen Concentration (FiO2) 41%.
  Interventions: Other: variable tidal volume ventilation (V-VCV)
- PRVC Group (Experimental): The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW), the upper limit of peak inspiratory pressure was 30 cmH2O, the maximum tidal volume (Vt_max) and the minimum tidal volume (Vt_min) was set at 10-20% of the base tidal volume (Vt_base). Respiratory Rate is 12, Inspiration to Expiration Ratio is 1:2, Positive End-Expiratory Pressure (PEEP) is 5cmH2O, and Inhaled Oxygen Concentration (FiO2) is 98%.
  Interventions: Other: pressure-regulated volume-controlled ventilation (PRVC)
- C-VCV Group (Experimental): The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW).The maximum tidal volume (Vt_max) and minimum tidal volume (Vt_min) were set at 10-20% of the basal tidal volume (Vt_base). Respiratory Rate 12. Inspiratory Flow Rate (IFR) 60L/min, Inspiratory to Expiratory Ratio (IER) 1:2, Positive End-Expiratory Pressure (PEEP) 5cm water column, and Inhaled Oxygen Concentration (FiO2) 98%.
  Interventions: Other: conventional volume-controlled ventilation (C-VCV)
- PCV Group (Experimental): The inspiratory pressure level is set, usually with an initial value of 20 cmH2O, a respiratory rate of 12, an inspiratory/expiratory ratio of 1:2, a positive end-expiratory pressure (PEEP) of 5 cm water column, and an inspired oxygen concentration (FiO2) of 98%.
  Interventions: Other: pressure-controlled ventilation (PCV)

INTERVENTIONS:
Other: variable tidal volume ventilation (V-VCV) — The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW).The maximum tidal volume (Vt_max) and minimum tidal volume (Vt_min) were set at 10-20% of the basal tidal volume (Vt_base). Respiratory Rate 12. Inspiratory Flow Rate (IFR) 60L/min, Inspiratory to Expiratory Ratio (IER) 1:2, Positive End-Expiratory Pressure (PEEP) 5cm water column, and Inhaled Oxygen Concentration (FiO2) 41%.
  Arms: V-VCV Group
Other: pressure-regulated volume-controlled ventilation (PRVC) — The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW), the upper limit of peak inspiratory pressure was 30 cmH2O, the maximum tidal volume (Vt_max) and the minimum tidal volume (Vt_min) was set at 10-20% of the base tidal volume (Vt_base). Respiratory Rate is 12, Inspiration to Expiration Ratio is 1:2, Positive End-Expiratory Pressure (PEEP) is 5cmH2O, and Inhaled Oxygen Concentration (FiO2) is 98%.
  Arms: PRVC Group
Other: conventional volume-controlled ventilation (C-VCV) — The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW).The maximum tidal volume (Vt_max) and minimum tidal volume (Vt_min) were set at 10-20% of the basal tidal volume (Vt_base). Respiratory Rate 12. Inspiratory Flow Rate (IFR) 60L/min, Inspiratory to Expiratory Ratio (IER) 1:2, Positive End-Expiratory Pressure (PEEP) 5cm water column, and Inhaled Oxygen Concentration (FiO2) 98%.
  Arms: C-VCV Group
Other: pressure-controlled ventilation (PCV) — The inspiratory pressure level is set, usually with an initial value of 20 cmH2O, a respiratory rate of 12, an inspiratory/expiratory ratio of 1:2, a positive end-expiratory pressure (PEEP) of 5 cm water column, and an inspired oxygen concentration (FiO2) of 98%.
  Arms: PCV Group

SUMMARY:
The purpose of this clinical trial was to understand the effects of variable tidal volume ventilation (V-VCV), pressure-regulated volume-controlled ventilation (PRVC), conventional volume-controlled ventilation (C-VCV), pressure-controlled ventilation (PCV), and open surgery (Open Surgery). controlled ventilation (C-VCV), pressure-regulated volume-controlled ventilation (PRVC), conventional volume-controlled ventilation (C-VCV), and pressure-controlled ventilation (PCV) for open surgery, video-assisted thoracoscopic surgery, and segmental lung resection. VATS), segmentectomy (Segmentectomy), lobectomy (Lobectomy), and pneumonectomy (Pneumonectomy) on oxygen saturation and pulmonary complications, and length of hospitalization.

The main question it aims to answer is: variable tidal volume ventilation (V-VCV), pressure-regulated volume-controlled ventilation (PRVC), conventional volume-controlled ventilation (C-VCV), and pressure-controlled ventilation (PCV).Does it decrease patient oxygen saturation, and does it increase pulmonary complications, length of hospitalization? Researchers compared variable tidal volume ventilation (V-VCV), pressure-regulated volume-controlled ventilation (PRVC), conventional volume-controlled ventilation (V-VCV), pressure-regulated volume-controlled ventilation (PRVC), conventional volume-controlled ventilation (C-VCV), and pressure-controlled ventilation (PCV) to compare them to see which mode of ventilation has the least physiologic disruption for the patient.

Participants will:

Select the appropriate surgical procedure according to the condition and be randomized to variable tidal volume ventilation (V-VCV), pressure-regulated volume-controlled ventilation (PRVC), conventional volume- controlled ventilation (C-VCV), pressure-controlled ventilation (PCV), and were checked after surgery.

Patients' oxygen saturation, pulmonary complications, length of hospitalization were recorded

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring any of open surgery, television-assisted thoracoscopic surgery (VATS), segmental lung resection (Segmentectomy), lobectomy, and total lung resection (Pneumonectomy).
* Patients who are able to receive any of the ventilation modes of controlled ventilation (C - VCV), pressure-regulated volume-controlled ventilation (PRVC), conventional volume-controlled ventilation (C - VCV), pressure-controlled ventilation (PCV), and variable tidal volume ventilation (V - VCV).

Exclusion Criteria:

* Patients with severe cardiac, hepatic, renal, and other vital organ dysfunction
* Patients with mental illness or cognitive disorders that prevent them from understanding the study and cooperating with the study process.
* Patients with hematologic disorders
* Pregnant or breastfeeding females

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
oxygen saturation | One week postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: January 2026-January 2036
Access Criteria: A proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed.